CLINICAL TRIAL: NCT01814306
Title: Comparison of the Effectiveness Between the LMA SupremeTM and the LMA ProsealTM for Airway Management in Patient Undergoing Elective Orthopaedic Surgery in Prone Position
Brief Title: Supreme LMA and Proseal LMA in Prone Anesthetized Patient
Acronym: SPLMA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Prince of Songkla University (Other)
Responsible Party: Principal Investigator, Chatchai Prechawai, Anesthesiology Department, Prince of Songkla University
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: SPLMA-100; SPLMA-100-CPrechawai (Registry Identifier: CPrechawai)
Record Dates: First submitted 2013-02-12; First posted 2013-03-19 (Estimated); Last update posted 2013-03-19 (Estimated); Status verified 2013-03

CONDITIONS: Inadequate or Impaired Breathing Pattern or Ventilation
Keywords: LMA Supreme,LMA Proseal,airway management,prone position
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Supreme (Active Comparator): Supreme LMA
  Interventions: Device: Supreme LMA
- Proseal (Active Comparator): Proseal LMA
  Interventions: Device: Proseal LMA

INTERVENTIONS:
Device: Supreme LMA — Use Supreme LMA to compare efficay with Proseal LMA in prone position insertion
  Arms: Supreme
Device: Proseal LMA — Use Proseal LMA to compare efficay with Supreme LMA in prone position insertion
  Arms: Proseal

SUMMARY:
There is no significant difference about success rate of two devices.

DETAILED DESCRIPTION:
There is no significant difference about success rate of two device: efficacy and safety

ELIGIBILITY:
Inclusion Criteria:

* American Society Anesthesiologists physical status I-III
* Patient undergo elective orthopedics surgery in prone position under general anaesthesia

Exclusion Criteria:

* Age <15year
* Non-fast
* Morbid obesity (BMI > 35kg/m2)
* Pregnancy
* Known or predicted difficult airway
* GERD
* History of laryngeal problem (injury,subglottic stenosis)
* Local pharyngeal problem (abscess,tumor)
* Poor dentation
* Pulmonary disease

Max Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2011-10; Primary Completion 2013-04 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
Success rate of insertion (quality of ventilation) | 1 year

SECONDARY OUTCOMES:
Ease of insertion, Complication and Glottic seal pressure | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Chatchai Prechawai, Study Chair — Prince of Songkla University
Locations (1):
- Faculty of Medicine, Prince of Songkla University, Hat Yai, Changwat Songkhla, Thailand